CLINICAL TRIAL: NCT04699968
Title: Phase II Clinical Trial of SHR-1701 With or Without Famitinib in the Treatment of Advanced or Metastatic NSCLC
Brief Title: A Trial of SHR-1701 With or Without Famitinib in Patients With Advanced or Metastatic NSCLC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor R & D Strategy Adjustment
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701-Ⅱ-206
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — SHR-1701

STUDY DESIGN:
Intervention Model Description: SHR-1701 with or without Famitinib
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: SHR-1701，Famitinib
- Treatment group B (Experimental)
  Interventions: Drug: SHR-1701

INTERVENTIONS:
Drug: SHR-1701，Famitinib — SHR -1701, Intravenous ；Famitinib, oral
  Arms: Treatment group A
Drug: SHR-1701 — SHR -1701, Intravenous
  Arms: Treatment group B

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of SHR-1701 with or without famitinib in patients with advanced or metastatic NSCLC

ELIGIBILITY:
Inclusion Criteria:

1. voluntarily participate in the study and sign the informed consent form;
2. 18 to 75 years old, both male and female;
3. histologically or cytologically confirmed stage IIIB-IV or recurrent NSCLC
4. one prior platinum-containing chemotherapy for advanced or metastatic disease;
5. measurable lesions by RECIST v1.1;
6. ECOG score: 0-1;
7. life expectancy ≥ 3 months;
8. adequate hematological, hepatic and renal function;
9. non-surgically sterile female subjects of childbearing age must have a negative serum HCG test.

Exclusion Criteria:

1. histologically or cytologically confirmed mixed SCLC and NSCLC;
2. known sensitising EGFR mutation and/or ALK translocation in patients with non-squamous NSCLC;
3. tumor infiltration into the great vessels on imaging;
4. active CNS metastases;
5. malignancies other than NSCLC within 5 years;
6. anticancer therapy within 4 weeks before the start of trial treatment;
7. persisting toxicity related to prior therapy of Grade > 1;
8. treatment with systemic immunostimulatory agents within 4 weeks;
9. treatment with systemic immunosuppressive agents within 2 weeks;
10. autoimmune diseases;
11. interstitial lung disease or other lung diseases that is symptomatic or may interfere the management of suspected drug-related pulmonary toxicity;
12. clinically significant cardiovascular or cerebrovascular diseases;
13. inadequately controlled hypertension;
14. history of hemoptysis (≥ 2.5mL of bright red blood per episode) within 1 month;
15. venous or arterial thrombosis within 6 months;
16. evidence of bleeding diathesis or coagulopathy;
17. use of anticoagulants or thrombolytic agents that has not been stable;
18. active Tuberculosis infection;
19. significant acute or chronic infections within 1 month;
20. known history of testing positive test for HIV or known AIDS;
21. hepatitis B virus or hepatitis C virus infection;
22. allergic to any component of the treatment regimen;
23. other conditions that in the opinion of the investigator would make participation in this clinical trial inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
ORR | determined by RECIST v1.1, up to approximately 1 year
  Objective Response Rate

SECONDARY OUTCOMES:
PFS | determined by RECIST v1.1, up to approximately 1 year
  Progression-Free-Survival
DCR | determined by RECIST v1.1, up to approximately 1 year
  Disease Control Rate
DoR | determined by RECIST v1.1, up to approximately 1 year
  Duration of Response
OS | up to approximately 1 year
  Overall Survival
AEs+ SAEs | determined by NCI-CTCAE V5.0, from the first drug administration to within 90 days for the last SHR-1701 dose
  Adverse Events and Serious Adverse Events